CLINICAL TRIAL: NCT07139353
Title: Linperlisib Combined With Chidamide in the Treatment of Relapsed or Refractory Peripheral T-cell Lymphoma: A Prospective, Multicenter, Open-label, Phase Ib/II Clinical Study
Brief Title: Linperlisib Combined With Chidamide in the Treatment of Relapsed or Refractory Peripheral T-cell Lymphoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, MD. PhD., Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-420
Record Dates: First submitted 2025-08-15; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Peripheral T Cells Lymphoma (PTCL)
MeSH Terms: interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Linperlisib Combined with Chidamide (Experimental): Patients will receive Chidamide 20 mg orally twice weekly (biw) in combination with Linperlisib at the RP2D (80 mg or 60 mg, po, qd). Each treatment cycle is 28 days.
  Interventions: Drug: Linperlisib; Drug: Chidamide

INTERVENTIONS:
Drug: Linperlisib — Linperlisib: 80 mg or 60 mg, po, qd (phase Ib); RP2D (phase II)
Drug: Chidamide — Chidamide: 20mg, po, biw

SUMMARY:
This is a prospective, multicenter, open-label, phase Ib/II clinical study to evaluate the safety and efficacy of linperlisib combined with chidamide in the treatment of relapsed or refractory peripheral T-cell lymphoma

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the clinical study; fully understand and be informed about the study and sign the Informed Consent Form (ICF); willing to comply with and capable of completing all trial procedures;
* Diagnosed with PTCL according to the 2022 revised WHO lymphoma classification standards based on pathological diagnosis by the research center
* Using the Lugano 2014 lymphoma efficacy evaluation criteria, the patient must have at least one measurable or evaluable lesion
* Treatment failure to at least one prior line of systemic standard therapy for PTCL.
* Age ≥ 18 years
* Expected survival greater than 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Adequate organ and bone marrow function

Exclusion Criteria:

* Accompanied by hemophagocytic lymphohistiocytosis (HLH)
* Lymphoma involvement in the central nervous system or meninges
* Active infections
* Uncontrolled clinical cardiac symptoms or diseases
* Currently using (or unable to stop at least one week prior to the first dose) a known CYP3A strong inducer or strong inhibitor.
* Currently using vitamin K antagonists, antiplatelet drugs, anticoagulants (or unable to stop them within one week prior to the start of the study treatment).
* History of Human Immunodeficiency Virus (HIV) infection and/or Acquired Immunodeficiency Syndrome (AIDS).
* Patients with mental disorders or those unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) for Phase 1b | The first cycle (each cycle is 28 days) after administration
  To identify the DLT
Overall response rate(ORR) for Phase 2 | Up to 24 months
  The proportion of patients who achieve complete remission (CR) or partial remission (PR) as the best response.

SECONDARY OUTCOMES:
Complete response rate (CRR) | Up to 24 months
  Defined as the proportion of patients who achieve complete remission as the best response
Duration of Response(DOR) | Up to 4 years
  To investigate the preliminary anti-tumor efficacy
Progression-free survival(PFS) | Up to 4 years
  To investigate the preliminary anti-tumor efficacy
Overall survival(OS) | Up to 4 years
  To investigate the preliminary anti-tumor efficacy

IPD SHARING:
Plan to Share IPD: Undecided